CLINICAL TRIAL: NCT04287153
Title: Evaluation of the Effectiveness of Cryotherapy in Slimming of the Abdomen and Saddlebags
Brief Title: Cryotherapy and Body Slimming
Acronym: Cryotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinic Cryo Esthetic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A01278-45
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Cryotherapy Effect; Weight Loss
Keywords: obesity; cryotherapy; weight loss; saddlebags
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Assessment of the effectiveness and tolerance of cryotherapy in the thinning of the abdomen and saddelbags
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Croytherapy on abdomen and saddlebags (Experimental): Six (6) to 10 applicators (application area of 17 cm X 6 cm) are applied on the dorsal side (back, waist, saddlebags) for 45 minutes and then on the ventral side (belly) for 45 minutes, with adjustments according to the size of the participant. The temperature applied with the device is variable (-10°c to -7°C).
  Interventions: Device: Cryotherapy on abdomen and saddlebags

INTERVENTIONS:
Device: Cryotherapy on abdomen and saddlebags — Application of variable temperature (-10°c to -7°c) on the treated areas using the cryotherapy device FG660L-006 (Beijing ADSS Development CO., Ltd)

SUMMARY:
The purpose of this study is to evaluate the efficacy of cryotherapy on the slimming of subcutaneous fat mass in the abdomen and saddlebags. Cryotherapy is a completely non-invasive method that induces a selective reduction of fat cells by localized and controlled cooling in areas such as the abdomen, flanks, inner knees, inner thighs, back and arms.

Adipose tissue is composed of two types of tissue: white and brown adipose tissue. Studies have shown that exposure to cold induces an increase in the number of brown adipocytes (detected by PET/CT-scan) under the effect of the hormone irisin produced by the muscles. In addition, another study has shown that prolonged exposure to cold reduces the size of brown adipocytes leading to thermogenesis, suggesting that cold exposure may contribute to the control of obesity.

The freezing technology of this cryotherapy unit allows the temperature of the subcutaneous adipose tissue to move almost instantaneously from -6°C to -10°C, gradually causing the reduction of subcutaneous adipose tissue.

DETAILED DESCRIPTION:
Prospective, monocentric pilot and comparative (before and after) study in simple blind (assessor different from the operator).

* The effectiveness of cryotherapy will be evaluated by the metric measurement of the treated areas: waist circumference, from the hips to the level of the saddlebags.
* Measurement of subcutaneous fat mass with iDXA scanner on treated areas
* Metabolic parameters from a blood test: Liver function (AST, ALT, gamma GT), inflammatory markers, plasmatic fatty acids, glycerol, total cholesterol, triglycerides, lipids, blood sugar, insulin, lactate.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old and non-menopausal with a BMI between 20 and 30 (20≥IMC≤30), with an overload of abdominal subcutaneous fat tissue and at the saddlebags

Exclusion Criteria:

* - < 18 years old.
* Pregnancy
* Breastfeeding
* Cold allergy: 2-minute ice cube test positive
* A waist/hip ratio indicative of a pathological fat distribution (>0.8 for women, >0.9 for men)
* Endocrine pathologies (Cushing's disease, endocrine tumours, unbalanced frank or labile hypothyroidism, hirsutism and hyper-androgenism, insulin resistance and/or unbalanced type 2 diabetes...)
* Neoplasia
* Psychiatric pathologies with or without treatment (Antidepressants, Neuroleptics, Anxiolytics...), well characterized anorexia-bulimia syndromes.
* Established alcoholism. Daily alcohol consumption should not exceed 2 glasses of wine per day.
* Digestive pathologies (especially hepatic) and functional digestive disorders (chronic constipation, alternating constipation-diarrhoea, chronic abdominal pain).
* Weaknesses of the abdominal wall (umbilical, inguinal, crural hernias)
* HIV in therapy
* Genetic deformities and diseases
* Vegetarian/vegetarian diet, macrobiotic diet
* Spasmophilia
* Surgery less than 3 months old
* Unbalanced coronary artery disease, untreated angina

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Metric measurements of the treated areas (cm) | 15 days after treatment
  The effectiveness of cryotherapy will be evaluated by the metric measurement of the treated areas: waist circumference, from the hips to the horse's breeches.
Metric measurements of the treated areas (cm) | 3 months after treatment
  The effectiveness of cryotherapy will be evaluated by the metric measurement of the treated areas: waist circumference, from the hips to the horse's breeches.

SECONDARY OUTCOMES:
iDXA scanner measurement | 15 days
  Measurement of subcutaneous fat mass in areas treated with the iDXA scanner
iDXA scanner measurement | 3 months
  Measurement of subcutaneous fat mass in areas treated with the iDXA scanner
Metabolic assessment | 15 days after treatment
  Metabolic assessment from a blood test: Liver function: Transaminase GOT, Transaminase GPT, Gamma GT (U/l)
Metabolic assessment | 15 days after treatment
  Total cholesterol, triglycerides, HDL cholesterol (g/l)
Metabolic assessment | 15 days after treatment
  Neopterin (nmol/l)
Metabolic assessment | 15 days after treatment
  leptin (pg/l)
Metabolic assessment | 15 days after treatment
  adipoleptin (mg/l)

CONTACTS AND LOCATIONS:
Overall Officials: Suva Loap, MD, Principal Investigator — Cryoesthetic
Locations (1):
- Cryoesthetic, Paris, France

REFERENCES:
- [Result] Aronne LJ. Epidemiology, morbidity, and treatment of overweight and obesity. J Clin Psychiatry. 2001;62 Suppl 23:13-22. PMID 11603881
- [Result] Kennedy J, Verne S, Griffith R, Falto-Aizpurua L, Nouri K. Non-invasive subcutaneous fat reduction: a review. J Eur Acad Dermatol Venereol. 2015 Sep;29(9):1679-88. doi: 10.1111/jdv.12994. Epub 2015 Feb 9. PMID 25664493
- [Result] Avram MM, Harry RS. Cryolipolysis for subcutaneous fat layer reduction. Lasers Surg Med. 2009 Dec;41(10):703-8. doi: 10.1002/lsm.20864. PMID 20014262
- [Result] Mulholland RS, Paul MD, Chalfoun C. Noninvasive body contouring with radiofrequency, ultrasound, cryolipolysis, and low-level laser therapy. Clin Plast Surg. 2011 Jul;38(3):503-20, vii-iii. doi: 10.1016/j.cps.2011.05.002. PMID 21824546
- [Result] Bernstein EF. Longitudinal evaluation of cryolipolysis efficacy: two case studies. J Cosmet Dermatol. 2013 Jun;12(2):149-52. doi: 10.1111/jocd.12036. PMID 23725309
- [Result] van der Lans AA, Wierts R, Vosselman MJ, Schrauwen P, Brans B, van Marken Lichtenbelt WD. Cold-activated brown adipose tissue in human adults: methodological issues. Am J Physiol Regul Integr Comp Physiol. 2014 Jul 15;307(2):R103-13. doi: 10.1152/ajpregu.00021.2014. PMID 24871967
- [Result] Lee P, Swarbrick MM, Ho KK. Brown adipose tissue in adult humans: a metabolic renaissance. Endocr Rev. 2013 Jun;34(3):413-38. doi: 10.1210/er.2012-1081. Epub 2013 Apr 2. PMID 23550082
- [Result] Manstein D, Laubach H, Watanabe K, Farinelli W, Zurakowski D, Anderson RR. Selective cryolysis: a novel method of non-invasive fat removal. Lasers Surg Med. 2008 Nov;40(9):595-604. doi: 10.1002/lsm.20719. PMID 18951424
- [Result] Zelickson B, Egbert BM, Preciado J, Allison J, Springer K, Rhoades RW, Manstein D. Cryolipolysis for noninvasive fat cell destruction: initial results from a pig model. Dermatol Surg. 2009 Oct;35(10):1462-70. doi: 10.1111/j.1524-4725.2009.01259.x. Epub 2009 Jul 13. PMID 19614940
- [Result] Coleman SR, Sachdeva K, Egbert BM, Preciado J, Allison J. Clinical efficacy of noninvasive cryolipolysis and its effects on peripheral nerves. Aesthetic Plast Surg. 2009 Jul;33(4):482-8. doi: 10.1007/s00266-008-9286-8. Epub 2009 Mar 19. PMID 19296153
- [Result] Dierickx CC, Mazer JM, Sand M, Koenig S, Arigon V. Safety, tolerance, and patient satisfaction with noninvasive cryolipolysis. Dermatol Surg. 2013 Aug;39(8):1209-16. doi: 10.1111/dsu.12238. Epub 2013 May 2. PMID 23639062
- [Result] Garibyan L, Sipprell WH 3rd, Jalian HR, Sakamoto FH, Avram M, Anderson RR. Three-dimensional volumetric quantification of fat loss following cryolipolysis. Lasers Surg Med. 2014 Feb;46(2):75-80. doi: 10.1002/lsm.22207. Epub 2013 Dec 3. PMID 24535759
- [Result] Saarelainen J, Hakulinen M, Rikkonen T, Kroger H, Tuppurainen M, Koivumaa-Honkanen H, Honkanen R, Hujo M, Jurvelin JS. Cross-Calibration of GE Healthcare Lunar Prodigy and iDXA Dual-Energy X-Ray Densitometers for Bone Mineral Measurements. J Osteoporos. 2016;2016:1424582. doi: 10.1155/2016/1424582. Epub 2016 Apr 27. PMID 27239366